CLINICAL TRIAL: NCT03836248
Title: Study of the Contribution of Osteopathic Treatment to Classic Medical Management in Patients With Chronic Low Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Pasteur (Other)
Responsible Party: Principal Investigator, Barthélémy de Truchis, Principal investigator, MD, Clinique Pasteur
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018-A00395-50; 2018-A00395-50 (Other: ID-RCB)
Record Dates: First submitted 2019-02-07; First posted 2019-02-11 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Chronic Low Back Pain
Keywords: Osteopathic treatment; Sham osteopathic treatment; Low back pain
MeSH Terms: conditions — Low Back Pain | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: Prospective monocentric study randomized into three parallel arms.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1-Current practice Medication treatment (Other): Medication treatment according to current practice.
  Interventions: Other: Current practice Medication treatment
- 2- Sham osteopathic treatment (Sham Comparator): Medication treatment according to current practice + sham osteopathic treatment.
  Interventions: Other: Sham osteopathic treatment; Other: Current practice Medication treatment
- 3- Osteopathic treatment (Experimental): Medication treatment according to current practice + osteopathic treatment.
  Interventions: Other: Osteopathic treatment; Other: Current practice Medication treatment

INTERVENTIONS:
Other: Osteopathic treatment — 5 osteopathic treatment sessions lasting 20 to 40 minutes. Each session include diagnosis according to the specific methodology "geometric model of osteopathy" and treatment of necessary elements and a control of osteopathic treatment at the end of the session.
  Arms: 3- Osteopathic treatment
Other: Sham osteopathic treatment — 5 sham osteopathic treatment sessions lasting 20 to 40 minutes. Each session include diagnosis according to the specific methodology "geometric model of osteopathy" and only contacts for no intent to treat. At the end of the session a control of the sham osteopathic treatment is performed.
  Arms: 2- Sham osteopathic treatment
Other: Current practice Medication treatment — Analgesic medication of level 1 or a combination of level 1 and 2. Acetaminophen 1 g x 3 / day Ibuprofen 400mg x 3 / day

SUMMARY:
The management of chronic low back pain is now part of a multi-disciplinary set of proposals with the aim of adapting for each patient orientations of both medicated and non-medicated care.

Very classically, analgesic treatment of stage I or II is of use, reinforced by the occasional use of NSAIDs in the absence of contraindication. In this medical attempt of the control of the pain associates a physical care (supervised exercises, physiotherapy care), cognitive and behavioral therapy, multidisciplinary care.

Osteopathic treatment is a specific manual diagnostic and therapeutic procedure.

This study aims to evaluate the relevance of providing osteopathic treatment in combination with classical medical treatment in the management of patients with chronic non-specific low back pain.

DETAILED DESCRIPTION:
The primary objective is to show that the addition of osteopathic treatment to classical medical treatment decreases pain for patients with chronic nonspecific low back pain.

This goal will be evaluated at 3 months by comparing

* the 3-month change in the level of pain observed in arm 3 (classical medical treatment + osteopathic treatment) versus that observed in arm 1 (classical medical treatment), and
* the 3-month change in the level of pain observed in arm 3 (classical medical treatment + osteopathic treatment) versus that observed in arm 2 (classical medical treatment+ sham osteopathic treatment ).

ELIGIBILITY:
Inclusion Criteria:

* Patient with chronic non-specific low back pain: degenerative lumbalgia and low back pain unrelated to anatomical lesions that have been evolving for more than 3 months.
* Patient affiliated with a social security scheme or equivalent
* Patient having signed the study informed consent form.

Exclusion Criteria:

* Patient with specific low back pain: patient with one of the following pathologies: degenerative neurological pathology; infectious pathology; fracture vertebral lesion less than 1 year; vertebral osteosynthesis material or canal narrowing.
* Patient following a treatment of the Morphinic or Neuroleptic type.
* Pregnant, breastfeeding or parturient woman
* Patient participating in another clinical study
* Protected patient: Major under some form of guardianship ; Hospitalized without consent

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 199 (Estimated)
Dates: Start 2019-10-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Pain VAS Visual Analog Scale | Change from baseline to 3 months
  The primary outcome is the change in the VAS score on a 0-100 mm scale between Day 0 (before the placement of any osteopathic manipulations for Arm 3 ( or sham osteopathic treatment for Arm 2) and J90 ( after the last osteopathic treatment session for Arm 3 (sham osteopathic treatment for Arm 2)).

SECONDARY OUTCOMES:
Pain VAS , level improvement | Baseline, Day 15, Month 1, Month 2, Month 3, Month 6
  The improvement of the pain level will be objectified by the measurement of the variation of the VAS score.
Relief Numerical scale | Day 15, Month 1, Month 2, Month 3, Month 6
  The intensity of relief will be objectified by measuring the variation of the "relief" score on a numerical scale. Numeric Scale Cotation between 0% (No Relief) to 100%(Full Relief)
Drug consumption | Baseline, Day 15, Month 1, Month 2, Month 3, Month 6
  Drug consumption will be collected by patients using a patient diary and converted to DDD ( Defined Daily Dose).
Hand-Ground Distance and Schöber test | Baseline, Day 15, Month 1, Month 2, Month 3, Month 6
  The efficacy of functional and quality of life therapies will be assessed through functional clinical examinations (Hand-Ground Distance and Schöber test )
Oswestry score | Baseline, Day 15, Month 1, Month 2, Month 3, Month 6
  The efficacy of functional and quality of life therapies will be assessed through the self questionnaire: the Oswestry questionnaire.
Adverse event | Day 15, Month 1, Month 2, Month 3, Month 6
  Adverse events will be collected and analyzed for each arm.
Elements of the osteopathic diagnosis | Day 1, Day 7, Day 15, Month 1 Month 2
  The elements of the osteopathic diagnosis will be collected by the treating osteopaths at the beginning and at the end of each treatment. Exploratory outcome, osteopathic diagnosis will be assessed by an internal osteopath questionnaire specifying anatomical localization of identified dysfunctions.

CONTACTS AND LOCATIONS:
Overall Officials: Barthélémy De Truchis de Varennes, MD, Principal Investigator — Clinique Pasteur; François Djabaku, DO, Study Chair; Barthélémy De Truchis de Varennes, MD, Study Chair — Clinique Pasteur
Locations (1):
- Clinique Pasteur, Toulouse, France

IPD SHARING:
Plan to Share IPD: No